CLINICAL TRIAL: NCT03793894
Title: Engaging Low SES Inpatient Smokers in LDCT Lung Cancer Screening: Enhanced Interventions That Include CHWs to Address SDH Barriers
Brief Title: Inpatient Smokers and LDCT Screening Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38353; LCD-507875 (Other Grant/Funding Number: American Lung Association (ALA))
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer Screening; Smoking Cessation
Keywords: Community health worker (CHW); Shared decision making (SDM); Low-dose computed tomography (LDCT)
MeSH Terms: conditions — Smoking Cessation | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care (Active Comparator): All trial participants will receive smoking cessation counseling (standard of care) and will be given the AHRQ "Is Lung Cancer Screening Right for me?" patient decision aid to review independently while in the hospital.
  Interventions: Behavioral: Smoking Cessation Counseling; Behavioral: Decision Aid
- Inpatient SDM + CHW Navigation (Experimental): In addition to the smoking cessation counseling and decision aid received by all subjects, intervention subjects will receive shared decision making (SDM) + CHW navigation.
  Interventions: Behavioral: Smoking Cessation Counseling; Behavioral: Decision Aid; Behavioral: Shared decision making (SDM); Behavioral: CHW Navigation

INTERVENTIONS:
Behavioral: Smoking Cessation Counseling — All participants will receive inpatient smoking cessation counseling by the tobacco-trained NP. Inpatient smoking cessation counseling is the standard of care at BMC.
Behavioral: Decision Aid — The AHRQ "Is Lung Cancer Screening Right for me?" patient decision aid is a 4-page paper format with the following features: 1) LDCT screening harms and benefits information, written in plain language and using pictographs, easily understood by those with low health literacy; 2) prompts to clarify patient values and preferences and to stimulate discussion about tradeoffs; 3) clear quit smoking messaging and resources (1-800-QUIT-NOW)
Behavioral: Shared decision making (SDM) — During the smoking cessation consultation, the nurse practitioner (NP) will conduct SDM, using the 4-page AHRQ "Is Lung Cancer Screening Right for me?" decision aid as a guide. The purpose of SDM is three-fold: 1) conduct a tailored discussion on tradeoffs of LDCT screening, consistent with Centers for Medicare & Medicaid Services (CMS) requirements for SDM using a decision aid; 2) directly connect interested patients to LDCT screening; 3) to empower and motivate patients to quit smoking within the LDCT screening context.
  Arms: Inpatient SDM + CHW Navigation
Behavioral: CHW Navigation — The CHW will meet with the participant after the SDM to initiate the coordination of outpatient tobacco treatment, referral to LCS, and resources to address the barriers to preventive services. The CHW will follow patients subjects in the intervention arm for 3 months to help navigate and address negative social determinants of health that are barriers to LCS and tobacco treatment. For patients who agree to screening, the CHW will schedule the appointment, arrange the transportation to appointment, and meet participant at the appointment to facilitate the screening.
  Arms: Inpatient SDM + CHW Navigation

SUMMARY:
Lung cancer suffers from large racial and socioeconomic disparities. Yet those at the highest risk of lung cancer death - current smokers, blacks, and individuals with low socioeconomic status (SES) and negative social determinants of health (SDH) - are less likely to receive preventive health services, including the two most effective interventions to reduce lung cancer mortality: tobacco dependence treatment and lung cancer screening (LCS) with low-dose computed tomography (LDCT). At Boston Medical Center (BMC) these preventive services are grossly underutilized, in part due to barriers our patients face in accessing these outpatient programs. Innovative approaches are needed to guide high-risk smokers to post-discharge early lung cancer detection services.

The overarching goal of this study is to reduce disparities in lung cancer morbidity and mortality by using hospitalization at an urban safety net hospital as an opportunity to connect high-risk smokers to both LDCT lung cancer screening and tobacco dependence treatment.

In addition to inpatient shared decision making [SDM] by an NP using a decision aid, screen-eligible smokers will also be connected with a community health worker (CHW) to facilitate access to outpatient smoking cessation counseling and LCS (CHW navigation).

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) among 128 hospitalized smokers at BMC (64 participants in each of two arms), to assess the effect of inpatient SDM + CHW Navigation (AHRQ LDCT screening decision aid + CHW + SDM discussion + smoking cessation counseling) compared to Enhanced Usual Care (smoking cessation counseling + decision aid) on LDCT screening completion at 3 months, patient knowledge, and smoking cessation at 6 months.

The research will meet two specific aims (SA1 and SA2).

SA1: To address barriers to engaging smokers in prevention and early detection of lung cancer, a pilot RCT (Pilot Study 2) will be conducted in which screen-eligible hospitalized smokers will be randomized to receive inpatient sdm + CHW navigation (inpatient SDM during smoking cessation counseling visits + CHW navigation to coordinate outpatient tobacco treatment, referral to LCS, and resources to address negative social determinant of health that present barriers to these preventive services) or Enhanced usual care (furnishing of LDCT screening decision aid during inpatient smoking cessation counseling visits). Compared to Enhanced Usual Care, it is hypothesized that inpatient sdm + CHW navigation will increase the number of patients completing LCS (1° outcome) and LCS knowledge, and biochemically validated smoking cessation at 6 months (2° outcome).

SA2: To collect stakeholder input to inform future implementation, Fifteen primary care providers (PCPs) will be interviewed to assess their impressions of the intervention, integration into workflow, and barriers to adoption. Fifteen smokers who received the intervention will be interviewed to learn their impressions of its utility and suggestions for improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized smoker at BMC
2. Meeting LDCT screening eligibility criteria: (age 55-80 years; ≥30-pack years smoking)
3. Current smoker (> 1 cigarette per day)
4. Able to speak, read, and understand English
5. Able and willing to comply with all study protocols and procedures
6. Having a PCP in the BMC network or one of the affiliated health centers

Exclusion Criteria:

1. Inability to tolerate surgical resection of a lung cancer, as defined by home oxygen therapy (an indicator of severe lung cancer or heart disease)
2. Active cancer (receiving treatment/new diagnosis) in prior 3 months or advanced stage cancer
3. Signs and symptoms of lung cancer or prior diagnosis of lung cancer
4. Already had chest CT (LDCT screening or other chest CT) in the past year
5. Pregnant

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
LDCT screening within 3 months post randomization | 3 months
  Data will be collected from the electronic health record (EHR) and the BMC lung cancer screening (LDCT) database.

SECONDARY OUTCOMES:
Knowledge of LDCT screening | baseline, 24 hours post enrollment
  Knowledge about LDCT screening will be measured with a 23-item instrument developed by Lau and colleagues and modified for a low health literacy population by Crothers. The instrument includes true/false and multiple choice questions that will be used to determine a total score representing knowledge of LDCT screening.
Self-report smoking cessation | 6 months
  Participants will be asked during telephone interview if they are smoking.
Biochemical validated smoking cessation | 6 months
  Participants who self-report quitting will be invited to complete the CO test for biochemical verification. This dichotomous outcome will be defined by biochemically verified 7-day point prevalence abstinence at 6 months. At study end, participants will be identified as smokers who 1) self-report abstinence, but are identified as smokers via biochemical validation (CO level >10 ppm), or 2) self-report abstinence, but refuse biochemical verification.

CONTACTS AND LOCATIONS:
Overall Officials: Hasmeena Kathuria, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kathuria H, Gunawan A, Spring M, Aijaz S, Cobb V, Fitzgerald C, Wakeman C, Howard J, Clancy M, Foreman AG, Truong V, Wong C, Steiling K, Lasser KE, Bulekova K, Wiener RS. Hospitalization as an opportunity to engage underserved individuals in shared decision-making for lung cancer screening: results from two randomized pilot trials. Cancer Causes Control. 2022 Nov;33(11):1373-1380. doi: 10.1007/s10552-022-01620-8. Epub 2022 Aug 23. PMID 35997854